CLINICAL TRIAL: NCT01381250
Title: Prediction and Treatment Outcome of Internet-based Treatment of Pathological Gambling With Three-year Follow-up
Brief Title: Effects of Internet-based Treatment of Pathological Gambling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Uppsala University (Other)
Responsible Party: The Swedish National Institute of Public Health, The Swedish National Institute of Public Health
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Spelstudie2
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2004-01

CONDITIONS: Pathological Gambling
Keywords: Pathological gambling according to DSM and having gambled at least once the past month.; Being atleast 18 years old
MeSH Terms: conditions — Gambling | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): The treatment was based on established cognitive behavior therapy methods, as described in self-help books (Hodgins, 2002; Ladouceur & Lachance, 2006). The text was divided into eight modules and was adapted for Internet use. The first four modules had a motivational interviewing focus and included building motivation for change by letting the participant answer open-ended questions that would evoke talk of change. The participants were encouraged to ask for input from their relatives on different aspects of their gambling. In addition, the first four modules included time line follow-back and mapping of the reasons for gambling. The remaining four modules were based on CBT. Each module included information and exercises and ended with three to eight essay-style questions. Feedback on homework assignments was usually given within 24 hr after participants had sent their answers via e-mail. Once weekly, a telephone call was made by the therapists to each participant.
  Interventions: Behavioral: cognitive behavior therapy

INTERVENTIONS:
Behavioral: cognitive behavior therapy — The treatment was based on established cognitive behavior therapy methods, as described in self-help books (Hodgins, 2002; Ladouceur & Lachance, 2006). The text was divided into eight modules and was adapted for Internet use. The first four modules had a motivational interviewing focus and included building motivation for change by letting the participant answer open-ended questions that would evoke talk of change. The participants were encouraged to ask for input from their relatives on different aspects of their gambling. In addition, the first four modules included time line follow-back and mapping of the reasons for gambling. The remaining four modules were based on CBT. Each module included information and exercises and ended with three to eight essay-style questions. Feedback on homework assignments was usually given within 24 hr after participants had sent their answers via e-mail. Once weekly, a telephone call was made by the therapists to each participant.

SUMMARY:
A trial testing the outcome of an Internet-based treatment of pathological gambling with the hypothesis that there will be improvements both immediately and up to 36 months. It is also hypnotized that treatment response can be predicted from background variables.

ELIGIBILITY:
Inclusion Criteria:

* Pathological gambling according to DSM and having gambled at least once the past month
* Being atleast 18 years old
* Living in Sweden

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2004-05; Primary Completion 2006-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The National Opinion Research Center DSM Screen for Gambling Problems (NODS) | 1 month

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | 1 week
Quality of Life Inventory | Present moment

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, PhD, Principal Investigator — Umeå University
Locations (1):
- University, Umeå, Sweden